CLINICAL TRIAL: NCT02859597
Title: Randomized. Controlled Trial of the Utilization of High Flow Nasal Cannula for Oxygenation of Sedated Morbidly Obese Patients in the Endoscopy Suite
Brief Title: Use of High Flow Nasal Cannula During Sedation of Morbidly Obese Patients in the Endoscopy Suite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-6677
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Morbid Obesity; Noninvasive Ventilation; Deep Sedation
MeSH Terms: conditions — Obesity, Morbid | interventions — Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- High Flow Nasal Cannula (Experimental): High flow nasal cannula will be utilized to deliver oxygen to morbidly obese patients undergoing deep sedation for gastrointestinal procedures.
  Interventions: Device: High flow nasal cannula
- Nasal Cannula (Active Comparator): Typical nasal cannula will be utilized to deliver oxygen to morbidly obese patients undergoing deep sedation for gastrointestinal procedures.
  Interventions: Device: Nasal Cannula

INTERVENTIONS:
Device: High flow nasal cannula — High flow nasal cannula at 50 liters per minute and 50% oxygen will initially be used for oxygenation.
  Arms: High Flow Nasal Cannula
Device: Nasal Cannula — Control group will receive oxygen via standard flow nasal cannula at 5 liters per minute (approximately an FiO2 of 0.35)
  Arms: Nasal Cannula

SUMMARY:
This study evaluates the ability of high flow nasal cannula versus nasal cannula to oxygenate morbidly obese patients undergoing moderate to deep sedation for gastrointestinal procedures.

DETAILED DESCRIPTION:
The respiratory physiology of morbidly obese patients is altered due to restriction of the chest wall motion which decreases pulmonary compliance. In addition, anatomical changes lead to an increased incidence of airway obstruction in morbidly obese patients during periods of sedation. Both a typical nasal cannula and high flow nasal cannula provide supplemental oxygen to the patients to prevent desaturation and hypoxia. However, the higher flow rates of high flow nasal cannulas are able to produce allows for washout of carbon dioxide from the respiratory system aiding with ventilation and creates 3 to 5 cm H2O of positive end expiration pressure which helps prevent collapse of the airway aiding with oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index greater than or equal to 40
* Scheduled for a gastrointestinal endoscopy that requires MAC sedation

Exclusion Criteria:

* Body Mass Index less than 40
* Pregnant
* Require either invasive or non-invasive ventilation for respiratory failure
* Use home oxygen
* Ventilation is via a tracheostomy
* The procedure is emergent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay S Berger, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berzin TM, Sanaka S, Barnett SR, Sundar E, Sepe PS, Jakubowski M, Pleskow DK, Chuttani R, Sawhney MS. A prospective assessment of sedation-related adverse events and patient and endoscopist satisfaction in ERCP with anesthesiologist-administered sedation. Gastrointest Endosc. 2011 Apr;73(4):710-7. doi: 10.1016/j.gie.2010.12.011. Epub 2011 Feb 12. PMID 21316669
- [Background] Nishimura M. High-Flow Nasal Cannula Oxygen Therapy in Adults: Physiological Benefits, Indication, Clinical Benefits, and Adverse Effects. Respir Care. 2016 Apr;61(4):529-41. doi: 10.4187/respcare.04577. PMID 27016353
- [Background] Corley A, Caruana LR, Barnett AG, Tronstad O, Fraser JF. Oxygen delivery through high-flow nasal cannulae increase end-expiratory lung volume and reduce respiratory rate in post-cardiac surgical patients. Br J Anaesth. 2011 Dec;107(6):998-1004. doi: 10.1093/bja/aer265. Epub 2011 Sep 9. PMID 21908497
- [Background] Kabon B, Nagele A, Reddy D, Eagon C, Fleshman JW, Sessler DI, Kurz A. Obesity decreases perioperative tissue oxygenation. Anesthesiology. 2004 Feb;100(2):274-80. doi: 10.1097/00000542-200402000-00015. PMID 14739800
- [Background] Standards of Practice Committee of the American Society for Gastrointestinal Endoscopy; Lichtenstein DR, Jagannath S, Baron TH, Anderson MA, Banerjee S, Dominitz JA, Fanelli RD, Gan SI, Harrison ME, Ikenberry SO, Shen B, Stewart L, Khan K, Vargo JJ. Sedation and anesthesia in GI endoscopy. Gastrointest Endosc. 2008 Nov;68(5):815-26. doi: 10.1016/j.gie.2008.09.029. No abstract available. PMID 18984096
- [Background] Rigg JD, Watt TC, Tweedle DE, Martin DF. Oxygen saturation during endoscopic retrograde cholangiopancreatography: a comparison of two protocols of oxygen administration. Gut. 1994 Mar;35(3):408-11. doi: 10.1136/gut.35.3.408. PMID 8150356

RESULTS

PARTICIPANT FLOW:
Groups:
- Nasal Cannula: Typical nasal cannula will be utilized to deliver oxygen to morbidly obese patients undergoing deep sedation for gastrointestinal procedures.
  High flow nasal cannula: High flow nasal cannula at 50 liters per minute and 50% oxygen will initially be used for oxygenation.
Period: Overall Study
Arm/Group | High Flow Nasal Cannula | Nasal Cannula
Started | 22 (started Dec 2016) | 19 (Started Dec 2016)
Completed | 22 (September 2018) | 19 (September 2018)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Flow Nasal Cannula | Nasal Cannula | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 19 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (12.5) | 43.4 (12.2) | 46 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Ability to Maintain Oxygenation
Description: The ease at which the Anesthesiologist is able to maintain adequate oxygenation during the period of sedation required for the procedure. the ability of each oxygen device to maintain oxygenation was based on the number of manipulations; more manipulations, the device is less effective at maintaining saturation for this population.
Time Frame: During the period of sedation, on average up to 1 hour
Measure: Mean (Standard Deviation); unit: manipulations
Groups:
- High Flow Nasal Canula: High flow nasal cannula will be utilized to deliver oxygen to morbidly obese patients undergoing deep sedation for gastrointestinal procedures.
  High flow nasal cannula: High flow nasal cannula at 50 liters per minute and 50% oxygen will initially be used for oxygenation.
- Nasal Canula: Typical nasal cannula will be utilized to deliver oxygen to morbidly obese patients undergoing deep sedation for gastrointestinal procedures.
  High flow nasal cannula: High flow nasal cannula at 50 liters per minute and 50% oxygen will initially be used for oxygenation.
Arm/Group | High Flow Nasal Canula | Nasal Canula
Number analyzed (Participants) | 22 | 19
manipulations | 0.55 (0.55) | 0.61 (1.03)

2. Secondary Outcome: Number of Participants Requiring Airway Adjuncts During Procedure
Description: The use of airway adjuncts such as oral and nasal airways to insure adequate oxygenation during procedure.
Time Frame: During the period of sedation, on average up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Nasal Cannula | Nasal Cannula
Number analyzed (Participants) | 22 | 19
Participants | 0 | 0

3. Secondary Outcome: Number of Participants Who Need an Increase in Fraction of Inspired Oxygen
Description: Need to increase the FiO2 to maintain adequate oxygenation
Time Frame: During period of sedation, on average up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Nasal Canula | Nasal Canula
Number analyzed (Participants) | 22 | 19
Participants | 6 | 3

ADVERSE EVENTS:
Time Frame: Subjects were observed up until their hospital discharge, on average up to 3 hours.
Arm/Group | High Flow Nasal Cannula | Nasal Cannula
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 0/22 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT02859597/Prot_SAP_000.pdf